CLINICAL TRIAL: NCT02003755
Title: The Effects of Continuous Passive Motion on Hypertonia of Soleus in Individuals With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Ya-Ju Chang, Professor, Chang Gung University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99-3614B
Record Dates: First submitted 2013-12-03; First posted 2013-12-06 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: Cerebral Palsy (CP)
Keywords: Cerebral palsy; Continuous passive motion; Hypertonia
MeSH Terms: conditions — Cerebral Palsy; Muscle Hypertonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Spastic CP (Experimental): continuous passive motion training
  Interventions: Procedure: Ankle continuous passive motion machine.

INTERVENTIONS:
Procedure: Ankle continuous passive motion machine. — A rehabilitation program of machine driven passive stretch.

SUMMARY:
Cerebral palsy (CP) is a group of disorders of the development of movement and posture but often changing motor impairment syndromes. The spastic subtypes are the most common manifestations of cerebral palsy who perform movement difficultly due to hypertonia. Decease of spinal cord pathway, hyperactivity of alpha and gamma motoneuron and reduction of presynaptic inhibition may cause tendon reflex increase and hypertonia in individuals with CP. There are many ways to improve the hypertonia. In the past studies, the fast repeated range of motion could reduce muscle's activation effectively. The polyarticular movement training might increase joint range of motion and reduce the muscle activation. But the polyarticular movement training is difficulty for some individuals with CP. The single joint movement training may achieve the same effect as the polyarticular movement training. The purpose of this study was to investigate the effects of continuation passive range of motion (CPM) training whether could get the improvement of soleus hypertonia in individuals with CP.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Spastic CP
* Modified Ashworth scale of Soleus > 1
* Ankle range of motion > 10 degrees

Exclusion Criteria:

* Fracture on lower Lower extremities
* BOTOX on ankle < 5 mouths

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2011-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Muscle tone tests | Baseline, 1, and 4 months.
  Measure of changes in Hypertonia measured by Modified Ashworth Scale (MAS).
Ankle range of motion | Baseline, 1, and 4 months.
  Measure of changes in Ankle range of motion.
Hoffman reflex (H-reflex) | Baseline, 1, and 4 months.
  Measure of changes in Hoffman reflex (H-reflex).

SECONDARY OUTCOMES:
Leg girth | Baseline,1 ,and 4 mouths.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan